CLINICAL TRIAL: NCT06929455
Title: Using Bitter Taste Receptor Blockers to Improve the Palatability of Pediatric Medicines: Trained Human Sensory Panels
Brief Title: Using Bitter Taste Receptor Blockers to Improve the Palatability of Pediatric Medicines
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Monell Chemical Senses Center (Other)
Collaborators: NIAID, Division of AIDS (contract funder) (Unknown); Advanced Biosciences Laboratories (ABL; primary contract holder) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 75N93024F00002; AI 75N93023D00001 (Other Grant/Funding Number: NIH NIAID)
Record Dates: First submitted 2025-04-07; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Healthy Adults
MeSH Terms: interventions — Flavoring Agents

STUDY DESIGN:
Intervention Model Description: There are no formal arms. Some samples will contain pharmaceutical ingredients without added flavors (control), and some samples will contain both pharmaceutical ingredients and flavor additives (experimental condition to determine if added flavors ingredients improve the flavor of the samples).
Masking Description: Samples for tasting will be presented with numeric identification codes (no verbal descriptors) and be presented in random order within a tasting session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- There are no study arms as typically defined in a clinical trial (Other): Various APIs will be presented with and without flavor additives. The list of APIs and additives will be developed as the study progresses, informed by ongoing work using in vitro taste assays. There are no formal, pre-specified study arms as typically defined in a clinical trial.
  Interventions: Other: Flavor additives

INTERVENTIONS:
Other: Flavor additives — Various flavors will be added to API samples. The particular APIs and flavor additives to be studied will be determined in part by on-going in work using in vitro taste models (cell systems expressing taste receptor proteins), so there is no full prespecified list.

SUMMARY:
Many people, particularly small children, must take drugs in liquid form because they cannot swallow pills or capsules. The bad taste of some liquid drugs can keep patients from taking drugs they need for their health. Our main goal in this research study is find ingredients that might make drugs taste better.

Participants in this research study will be healthy adults between the ages of 18 and 60 years old. Participants will taste samples (liquids or gels) containing active pharmaceutical ingredients (substances in medications that produce desired health effects). After tasting each sample participants will spit out the sample and rinse with water (no samples will be swallowed). Active pharmaceutical ingredients of current interest are: 1) tenofovir alafenamide, used to treat HIV infection and hepatitis B, 2) rifampicin, used to treat tuberculosis, 3) rifapentine, used to treat tuberculosis, and 4) levofloxacin, used to treat various bacterial infections). Other active pharmaceutical ingredients may be added as the study goes forward. Participants will be instructed to taste samples both with and without experimental flavor ingredients added and judge how the samples taste. People who volunteer for the study will be instructed to complete many repeated visits to the Monell Center (University City area of Philadelphia) for tasting sessions. Tasting visits will last between 1 and 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 60;
* Generally healthy by self-report;
* All races/ethnicities, both men and women;
* Able to provide informed consent;
* Able to attend repeated visits to Monell for sensory testing;
* Willing to follow instructions (e.g., refrain from eating or drinking for at least 1 hour before sessions, willing to remain on site for one hour after tasting an API that the participant has never tasted before). -

Exclusion Criteria:

* Under 18 or over 60;
* Pregnant, nursing, or plans to become pregnant;
* Unable to provide consent (including limited ability to understand written and spoken English);
* Tobacco, vape, marijuana, or tetrahydrocannabinol cartridge users. We will accept people who have used tobacco or marijuana products on occasion, but not regular users;
* Known drug or food allergies of any kind;
* Diabetes or other metabolic disorder;
* Liver issues of any kind, including viral hepatitis;
* Kidney issues of any kind;
* Other chronic illness, including cardiovascular, neurological, immune disorders, or any other serious acute or chronic condition
* Dentures or other major dental implants;
* Condition affecting the oral cavity, including dry mouth, burning mouth syndrome, active sores or blisters, geographic tongue, or other disorders
* Current infection or cold, flu, or infection with SARS-CoV-2 within the last four weeks;
* Unable to taste or smell
* Daily use, or use within the last four weeks, of either prescription or over-the-counter medications (except for birth control)
* History of tuberculosis (including latent tuberculosis), positive skin or other tuberculosis test at any time in the past, birth in or residence in a country with high tuberculosis rates, known contact with someone who is tuberculosis positive
* HIV infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Ratings of flavor intensity | Through study completion, between about 2 months and 3 years, depending on the number of API-flavor combinations individual participants choose to evaluate
  Ratings of oral sensation (e.g., bitterness, sourness, astringency, etc.) made using the general Labeled Magnitude Scale. Values range from 0 (no sensation) to 100 (strongest imaginable sensation)

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Wise, Ph.D., Principal Investigator — Monell Chemical Senses Center
Locations (1):
- Monell Chemical Senses Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with qualified researchers upon request, and may be made available in managed repositories as allowed by funder and journal policy.
Time Frame: De-identified data will be made available upon publication of results, as consistent with applicable Journal policies. Once available, data will be available indefinitely. Note, however, that individual participants will have the option to opt out of the data-base upon request to the study PI. Once such a request is received, data for the individual participant concerned will no longer be available.
Access Criteria: Data will be made available to qualified researchers by the study PI upon request (after publication). If data are placed in managed repositories (e.g., NIH-run managed repository), qualifications will be determined by the managers of the repository

DOCUMENTS (1):
  • Informed Consent Form (2025-02-28): https://cdn.clinicaltrials.gov/large-docs/55/NCT06929455/ICF_000.pdf